CLINICAL TRIAL: NCT05747183
Title: Comparison of Post Endodontic Pain for Preparation Using ProTaper Gold and ProTaper Ultimate Systems. A Randomized Clinical Study
Brief Title: Effect of ProTaper Ultimate System on Post-endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Principal Investigator, Rania Zaarour, Assistant Professor of Cell Biology and Researcher, Gulf Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB/COD/STD/33/June-2022
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Post Endodontic Pain
Keywords: Post endodontic pain; ProTaper Gold; ProTaper Ultimate; Root canal preparation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProTaper Ultimate (Experimental): Root canal preparation using ProTaper Ultimate files.
  Interventions: Procedure: ProTaper Ultimate
- ProTaper Gold files (Active Comparator): Root canal preparation using ProTaper Gold files.
  Interventions: Procedure: ProTaper Gold

INTERVENTIONS:
Procedure: ProTaper Ultimate — Root canal preparation using ProTaper Ultimate files.
  Arms: ProTaper Ultimate
Procedure: ProTaper Gold — Root canal preparation using ProTaper Gold files.
  Arms: ProTaper Gold files

SUMMARY:
This clinical trial aims to compare the effect of Pro Taper Ultimate and Pro Taper Gold files on post-endodontic pain in molars with symptomatic apical periodontitis.

The main question it aims to answer is:

If there is a difference in post-endodontic pain intensity following root canal preparation using Pro Taper Ultimate and Pro Taper Gold files in molar diagnosed with symptomatic apical periodontitis?

Participants will undergo root canal treatment using Pro Taper Ultimate and Pro Taper Gold files.

Researchers will compare [Pro Taper Ultimate and Pro Taper Gold files] to see the intensity of post-endodontic pain

DETAILED DESCRIPTION:
The study will be conducted on 40 first mandibular molars; with 20 first mandibular molars in each group (n=20). The patient will be asked to pick an opaque sealed envelope that will contain a number from 1 to 2. The resultant number will determine in which group the participants will be placed.

Group I: Root canal preparation using Pro Taper Ultimate. Group II: Root canal preparation using Pro Taper Gold.

Procedural steps:

1. Vitality will be assessed using cold tests and electric pulp testing before the procedure is carried out. Besides, mobility, palpation, and percussion tests will be done to assess periapical health. In order to ensure that the cold and electrical pulp tests are working, and a response is elicited, both tests will be carried out on patients not included in the study.
2. All the patients will receive local anesthesia: 2% lidocaine with 1:100,000 epinephrine.
3. Each tooth will be isolated using a rubber dam, and the access cavity will be prepared using a round bur (no.4) and tapered fissure diamond bur under copious water.
4. After removal of coronal pulp tissues using a sterile excavator, the working length will be determined with stainless steel hand K-files size #10 and the use of an apex locator and confirmed using intraoral periapical radiographs.
5. Hand instrumentation to 15-size K files.
6. Group I will be prepared using ProTaper Ultimate files.
7. Group II will be prepared using ProTaper Gold files.
8. Apical patency will be maintained throughout the shaping procedure using the #10 file between each instrument.
9. All the canals will be irrigated with 10 mL of 3% NaOCl between each file during the whole preparation procedure.
10. All the root canals will be obturated directly after preparation.
11. All the teeth will be restored using resin composite restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patient was diagnosed with symptomatic irreversible pulpits and symptomatic apical periodontitis.
* 18-70 years old patients
* Permanent mandibular first molars.
* Teeth with a fully matured root.
* Restorable teeth indicated for endodontic treatment.
* Healthy patients.

Exclusion Criteria:

* Complex root canal morphology
* Calcified roots.
* Teeth with internal and external resorption.
* Medically compromised patients.
* Restricted mouth openings (trismus).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The level of post-endodontic pain | 24 hours
  Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be)
The level of post-endodontic pain | 72 hours
  Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be)
The level of post-endodontic pain | 1 week
  Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be)

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates

REFERENCES:
- [Derived] Hajwel M, Elemam R, Elsewify T, Eid B. Effect of ProTaper Ultimate and ProTaper Gold on Postoperative Pain in Mandibular First Molars With Symptomatic Irreversible Pulpitis and Symptomatic Apical Periodontitis: A Randomized Control Clinical Trial. Pain Res Manag. 2025 Oct 30;2025:9718875. doi: 10.1155/prm/9718875. eCollection 2025. PMID 41211526